CLINICAL TRIAL: NCT04363905
Title: Supplemental Iron Improves Submaximal Exercise Performance in Non-anemic Iron Depleted Mexican Women: A Randomized Placebo Control Trial
Brief Title: Supplemental Iron Improves Submaximal Exercise Performance in Non-anemic Iron Depleted Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 012002
Record Dates: First submitted 2019-10-11; First posted 2020-04-27 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency (Without Anemia)
Keywords: iron deficient non-anemic; supplementation; randomized control trial; submaximal intermittent exercise; serum ferritin; body iron
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 100 mg lactose capsule
  Interventions: Dietary Supplement: Placebo
- Ferrous sulfate (Experimental): 20 mg ferrous sulfate and lactose capsule
  Interventions: Dietary Supplement: Ferrous sulfate

INTERVENTIONS:
Dietary Supplement: Placebo — 100 mg lactose per day for 6 weeks
  Arms: Placebo
Dietary Supplement: Ferrous sulfate — 20 mg per day of elemental iron for 6 weeks
  Arms: Ferrous sulfate

SUMMARY:
The specific aims of the current study were: 1) To determine the prevalence of IDNA in a sample of Mexican women of reproductive age and 2) To determine how iron supplementation in IDNA women influences physical work capacity during submaximal exercise . The researchers hypothesized that marginally iron depleted women will have improved physical work capacity during submaximal intermittent exercise tests after dietary iron supplementation. However, no improvement in peak maximal oxygen consumption after dietary iron supplementation because they will remain non-anemic.

DETAILED DESCRIPTION:
Recent estimates of the prevalence of anemia among non-pregnant Mexican women of reproductive age range from 15 percent for a nationally representative sample from the 1988 National Nutrition Survey to 29 percent for low socioeconomic women from the PROGRESA baseline survey of 1998 (Mexican Ministry of Health, unpublished report). The cause of most of this anemia is iron deficiency. It can be assumed that time between 15 and 30 percent of Mexican women also experience iron deficiency without also experiencing anemia. In some studies of anemic women, iron deficiency has been shown to result in reduced physical performance as measured by VO2max (the oxygen consumption at maximum physical exertion), presumably due to reduced oxygen (02) transport related to the reduced hemoglobin (Hb) concentration. However, no effects of iron deficiency have been shown on VO2max in women who were not anemic. Given that Hb concentration is not reduced in iron deficient non anemic women, it is expected that VO2max remains unaffected. However, this less severe form of iron deficiency may still affect physical performance. The important role of iron in the synthesis of many of the enzymes involved in oxidative metabolism suggests that moderate levels of iron deficiency may impair muscular energy transformation at levels of exertion that are not as severe as those reflected in VO2max. The choice of the appropriate sub maximal physical performance test is therefore critical to successful demonstration of the effects of moderate iron deficiency on response to exercise stress.

In this study the investigators proposed to test the effects of iron deficiency on physical performance using a randomized double blind design that assigns marginally iron depleted, physically active women between 18 and 45 years to two treatments. One half of the women will be randomly assigned to a group that receives a daily oral iron supplement (20 mg of elemental iron as slow release ferrous sulfate) while the remaining women received a placebo. Investigators anticipated that iron supplementation would replete iron body stores in all women and increase Hb only in those who are marginally anemic. Investigators tested the physical performance response to iron treatment with two exercise tests. It was hypothesized that VO2max would not be affected by iron supplementation. A graded submaximal exertion test (30 60% of VO2max) to estimate energy expenditure (EE), gross efficiency (GE), and net efficiency (NE) was administered to test for an increase in work efficiency due to iron supplementation.

This study has important implications for the definition of dietary iron requirements in this segment of the Mexican population. The physical performance test used in this study (EE, GE, and NE), while well recognized, have never been applied to this type of research question nor has it been examined in relation to endurance performance in Mexican women. Investigators believe that previous reliance on the VO2max test to measure performance has biased conclusions toward concern only for the anemic subject, while the less severe forms of iron deficiency have been considered benign.

This study, if successful in supporting the stated hypotheses, will serve as further confirm the deleterious effects of iron deficiency without anemia and justify future research on more practical measures of performance related to female economic productivity and time and effort allocated to child care and household responsibilities.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking

Exclusion Criteria:

* acute or chronic injury or illness at time of screening, hemolytic anemia
* physician-diagnosed asthma, musculoskeletal problems, or eating disorders
* pregnant or lactating, pregnant with the previous year
* excessive alcohol consumption or recent use of recreational drugs
* recent history of eating disorders, or use of prescription medications and/or vitamin or mineral supplements that would interfere with dietary iron absorption

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2000-04-01 (Actual); Primary Completion 2000-08-31 (Actual); Study Completion 2000-12-31 (Actual)

PRIMARY OUTCOMES:
Marker of iron status: Hemoglobin | 6 weeks
  g/L
Marker of iron status: serum ferritin | 6 weeks
  ug/L
Marker of iron status: serum transferrin receptor | 6 weeks
  mg/L
Marker of iron status: serum iron | 6 weeks
  umol/L
Marker of iron status: total iron binding capacity | 6 weeks
  umol/L
Marker of iron status: transferrin saturation | 6 weeks

SECONDARY OUTCOMES:
Physical performance | 6 weeks
  Submaximal and maximal cycling ergometry was used to assess physical performance
Fatigue resistance | 6 weeks
  Maximal voluntary static contractions (MVCs) with dynamic knee extensions was used to assess fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Jere D Haas, PhD, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

REFERENCES:
- [Background] Brutsaert TD, Hernandez-Cordero S, Rivera J, Viola T, Hughes G, Haas JD. Iron supplementation improves progressive fatigue resistance during dynamic knee extensor exercise in iron-depleted, nonanemic women. Am J Clin Nutr. 2003 Feb;77(2):441-8. doi: 10.1093/ajcn/77.2.441. PMID 12540406